CLINICAL TRIAL: NCT05085821
Title: Cardio-visual Stimulation in Augmented Reality for Pain Reduction
Acronym: HEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Union de Gestion des Etablissements des Caisses d'Assurance Maladie - Nord Est (Other)
Collaborators: Mindmaze SA (Industry)
Responsible Party: Principal Investigator, Amélie Touillet, Principal Investigator, Union de Gestion des Etablissements des Caisses d'Assurance Maladie - Nord Est
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRR-CLP-2019-4
Record Dates: First submitted 2021-05-03; First posted 2021-10-20 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2022-12

CONDITIONS: Regional Pain Syndrome; Chronic Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental 1: HEART - Placebo - HEART - Placebo (Experimental): The patient receives visual feedback in an augmented reality environment in four session, over two weeks.
  Week 1: HEART, Placebo (after >24hour washout) Week 2: HEART, Placebo (after >24hour washout)
  Interventions: Device: HEART; Device: Placebo
- Experimental 2: HEART - Placebo - Placebo - HEART (Experimental): The patient receives visual feedback in an augmented reality environment in four session, over two weeks.
  Week 1: HEART, Placebo (after >24hour washout) Week 2: Placebo, HEART (after >24hour washout)
  Interventions: Device: HEART; Device: Placebo
- Experimental 3: Placebo - HEART - Placebo - HEART (Experimental): The patient receives visual feedback in an augmented reality environment in four session, over two weeks.
  Week 1: Placebo, HEART (after >24hour washout) Week 2: Placebo, HEART (after >24hour washout)
  Interventions: Device: HEART; Device: Placebo
- Experimental 4: Placebo - HEART - HEART - Placebo (Experimental): The patient receives visual feedback in an augmented reality environment in four session, over two weeks.
  Week 1: HEART, Placebo (after >24hour washout) Week 2: Placebo, HEART (after >24hour washout)
  Interventions: Device: HEART; Device: Placebo

INTERVENTIONS:
Device: HEART — In an augmented reality environment, the patient receives visual feedback in synchrony with their cardiac-cycle (HEART)
Device: Placebo — In an augmented reality environment, the patient receives visual feedback out-of-synchrony with their cardiac cycle (Placebo)

SUMMARY:
The objective of this study is to evaluate the feasibility and efficacy of an Augmented Reality (AR) biofeedback intervention to alleviate pain symptoms in individuals suffering from chronic pain of the hand and/or the forearm.

DETAILED DESCRIPTION:
Chronic pain is a major public health problem with implications for high health care costs, lost productivity and an estimated financial burden of $500 billion. Individuals with chronic pain are also at an increased risk of developing an opioid use disorder.

Chronic pain has previously been associated with a distorted body representation, in particular of the affected body parts. Virtual Reality (VR) studies using embodiment-, respiration-, and heart-beat related feedback have demonstrated positive effects for induced pain in healthy participants (e.g., increased pain thresholds) and chronic pain in patient populations (e.g., decreased subjective pain, improved functionality, improved physiological markers of pain). Based on these studies, the AR intervention evaluated here aims to alleviate subjective pain symptoms and improve physiological pain markers in chronic pain patients using heartbeat-related feedback.

This within-subject study will compare subjective pain ratings before, during, and after an AR intervention that provides visual feedback of participants' on-going heartbeat in relation to their affected limb. Primary outcomes include subjective reports from participants (perceived efficacy, acceptability, and demand) and the intervention's clinical feasibility, including reports from therapists. Secondary outcomes include changes in heart rate and variability.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years of age
* Present permanent chronic pain (for more than 3 months), secondary to a peripheral pathology (traumatic, orthopedic or neurological), located in the hand or forearm.

Exclusion Criteria:

* Pregnant women
* People in emergency situations
* Persons unable to give informed consent
* Persons who are mentally or linguistically unable to understand the research test instructions
* Individuals who are not available to complete the entire study protocol
* Cognitive impairments that prevent the use of the equipment
* Psychiatric disorders
* Patients with seizure disorders
* Patients with central hemineglect
* Pain secondary to central nervous system pathology
* Patients with arrhythmia
* Patients with head tremors or head shaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Change in perceived pain | change in pain rating will be evaluated when participants first wear the Head-Mounted Display (baseline), after 3 minutes of video-passthrough (Pre), after 3 minutes of cardio-visual stimulation (post), after 3 minutes of video-passthrough (final)
  The patient moves a cursor on a Visual Analog Scale to indicate their currently perceived level of pain. The gauge ranges from "no pain" (0) to "worst pain imaginable" (10).
Change in Heart-Rate Variability (time domain) | a change in heart-rate variability will be evaluated between baseline (pre), intervention, and immediately following intervention (post)
  time-domain metrics of heart-rate variability [ms]
Change in Heart-Rate Variability (frequency domain) | a change in heart-rate variability will be evaluated between baseline (pre), intervention, and immediately following intervention (post)
  frequency-domain metric of heart-rate variability (power)

SECONDARY OUTCOMES:
Questionnaire | The first day of the study
  Questionnaire on the sensations, usability, and satisfaction with the augmented reality stimulation using a Visual Analog Scale (0-10) where higher scores indicate agreement with the questionnaire item.
Questionnaire | The second day of the study
  Questionnaire on the sensations, usability, and satisfaction with the augmented reality stimulation using a Visual Analog Scale (0-10) where higher scores indicate agreement with the questionnaire item.
Questionnaire | The third day of the study
  Questionnaire on the sensations, usability, and satisfaction with the augmented reality stimulation using a Visual Analog Scale (0-10) where higher scores indicate agreement with the questionnaire item.
Questionnaire | The fourth day of the study
  Questionnaire on the sensations, usability, and satisfaction with the augmented reality stimulation using a Visual Analog Scale (0-10) where higher scores indicate agreement with the questionnaire item.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Paysant, Pr, Principal Investigator — UGECAM Nord Est
Locations (1):
- Institut Régional de Médecine Physique et de Réadaptation, Nancy, France